CLINICAL TRIAL: NCT03981718
Title: Adipose-Induced Regeneration of Breast Skin (AIR Breast) to Treat Post-Mastectomy Radiation Injury in Breast Cancer Patients: A Randomized, Prospective Pilot Study
Brief Title: Adipose-Induced Regeneration of Breast Skin to Treat Post-Mastectomy Radiation Injury in Breast Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low/slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-002792; NCI-2022-11026 (Registry Identifier: NCI)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group: Standard (Active Comparator): Breast cancer subjects with current injury to irradiated skin at the post-mastectomy site will receive fat grafting procedure per standard of care during their 2nd stage breast reconstruction.
  Interventions: Procedure: Fat grafting
- Group: Experimental (Experimental): Breast cancer subjects with current injury to irradiated skin at the post-mastectomy site will receive their fat grafting procedure until 6 months after their 2nd stage breast reconstruction.
  Interventions: Procedure: Fat grafting

INTERVENTIONS:
Procedure: Fat grafting — Lipoaspirates will be collected from the own subjects abdominal fat tissue, during the 2nd stage breast reconstruction and will be injected on each affected breast during the insertion of the permanent breast implant in the 2nd stage of breast reconstruction

SUMMARY:
Researchers are trying to identify the therapeutic effect of injection into the subcutaneous tissue to treat radiation-induced skin injury of post mastectomy in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females above 18 years old
* Diagnosis with breast cancer, who will be treated by mastectomy and undergo radiotherapy, and will receive breast reconstruction
* Able and willing to sign consent to participate

Exclusion Criteria:

* Breast cancer patients that do not accept to participate
* Patients with previous breast reconstruction surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Increase in skin quality | 18 months
  Number of subjects to show reverse radiation-induced skin injury
Physical Well-Being Using the BREAST-Q Reconstruction Module | 12 months, 18 months
  Change in BREAST-Q patient-reported questionnaire to assess quality of life and patient satisfaction by using questions pertaining to the function and participation in activities after fat grafting. Subjects are asked to answer 16 questions on how often they experienced each symptom, using a score of 1 to 5, where 1 was none of the time and 5 was very often. Answers from these questions were combined to provide a total physical well-being score (for a total possible range of 16-80). Lower scores reflected fewer symptoms and higher satisfaction where higher scores reflected more symptoms and less satisfaction.
Effects of skin disease on quality of life | 12 months, 18 months
  Change in patient-reported Skin-16 questionnaire used to assess skin condition after fat grafting by using 16 questions on how often subjects skin condition has bothered them during the past week, using a score of 0 to 6, where 0 is never bothered and 10 is always bothered.
Skin Toxicity Costs | 12 months, 18 months
  Change in patient-reported skin toxicity costs questionnaire used to assess the economic impact of skin changes due to radiation after fat grafting by using 7 questions asking subjects to report total costs and itemized spending on specific items related to post procedure care.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Forte, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials